CLINICAL TRIAL: NCT06036927
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Clinical Trial to Evaluate the Efficacy, Safety and Pharmacokinetics of TQC2731 Injection in the Treatment of Chronic Sinusitis With Nasal Polyps.
Brief Title: A Clinical Study of TQC2731 Injection in the Treatment of Chronic Rhinosinusitis With Nasal Polyps
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQC2731-II-02
Record Dates: First submitted 2023-09-01; First posted 2023-09-14 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-03

CONDITIONS: Chronic Sinusitis; Nasal Polyps
MeSH Terms: conditions — Nasal Polyps

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TQC2731 injection 210 mg (Experimental): TQC2731 injection 210 mg combined with Mometasone Furoate Aqueous Nasal Spray, 28 days as a treatment cycle.
  Interventions: Drug: TQC2731 injection
- TQC2731 injection 420 mg (Experimental): TQC2731 injection 420 mg combined with Mometasone Furoate Aqueous Nasal Spray, 28 days as a treatment cycle.
  Interventions: Drug: TQC2731 injection
- TQC2731 matching placebo (Placebo Comparator): TQC2731 matching placebo combined with Mometasone Furoate Aqueous Nasal Spray, 28 days as a treatment cycle.
  Interventions: Drug: TQC2731 matching placebo

INTERVENTIONS:
Drug: TQC2731 injection — TQC2731 injection is a thymic stromal lymphopoietin (TSLP) monoclonal antibody.
  Arms: TQC2731 injection 210 mg; TQC2731 injection 420 mg
Drug: TQC2731 matching placebo — It'a a placebo injection without active substances.
  Arms: TQC2731 matching placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled Phase II clinical trial to evaluate the efficacy, safety and pharmacokinetics of TQC2731 injection in the treatment of Chronic Sinusitis with Nasal Polyps.

ELIGIBILITY:
Inclusion Criteria:

* Subjects sign informed consent before study, fully understand the purpose, procedures and possible adverse reactions of the study;
* Male and female, ≥18 years old and ≤ 75 years old;
* Bilateral chronic rhinosinusitis with nasal polyps (CRSwNP) who met the diagnostic criteria of the Chinese Guidelines for the Diagnosis and Treatment of chronic rhinosinusitis (2018);
* Received nasal polyp surgery or received systemic glucocorticoid treatment 2 years before screening;
* Bilateral nasal polyp score (NPS) ≥5 and each nostril was scored ≥ 2 when screening and randomization;
* Nasal congestion score (NCS) ≥2 when screening and randomization;
* Persistent nasal leakage or smell decrease or loss last more than 8 weeks before screening;
* Sinonasal outcome testing 22 (SNOT-22) score ≥ 30 when screening and randomization;
* Subjects received steady dose of intranasal glucocorticoids (INCS) over 4 weeks before screening (subjects agree use Mometasone Furoate Aqueous Nasal Spray (MFNS) while studying);
* Subjects with asthma start inhaled stable dose of glucocorticoid therapy over 4 weeks before screening, and are willing to keep the dose during whole study;
* MFNS medication compliance ≥70%, subjects daily symptom assessment compliance ≥70% through Patient dairy;
* Subjects agree to take effective non-pharmaceutical contraception from signing informed consent to 6 mouth after last administration.

Exclusion Criteria:

* Presence of conditions/concomitant diseases that affect the evaluation of efficacy, such as:

  1. Posterior nostril polyps;
  2. Deviation of the nasal septum resulted in obstruction of at least one nostril;
  3. Acute sinusitis, nasal infection, or upper respiratory tract infection had occurred 2 weeks before screening, screening period or mediation period;
  4. Drug induced rhinitis;
  5. Allergic granulomatous vasculitis (Churg-Strauss syndrome), granuloma with poly vasculitis (Wegener's granuloma), Young syndrome, Kartagener syndrome, or other dysphoric ciliary syndrome, with cystic fibrosis;
  6. Imaging suspected or confirmed fungal sinusitis;
  7. NPS cannot be evaluated due to nasal surgery to alter the structure of the lateral nasal wall;
  8. Subjects with nasal malignancies and benign tumors (papilloma, blood furuncle, etc.)
* Any type of active malignancy or a history of malignancy (Patient with basal cell carcinoma, skin localized squamous cell carcinoma or carcinoma in situ of cervix, can participate in the study if curative treatment was completed for more than 12 months prior to visit 1; Patients with other malignant tumors can participate in the study if curative therapy had been completed for at least 5 years prior to visit 1);
* Active autoimmune disease (including but not limited to Hashimoto's thyroiditis, Graves disease, Inflammatory bowel disease, Primary biliary cholangitis, Systemic lupus erythematosus, Multiple sclerosis and other neuroinflammatory diseases, Psoriasis vulgaris, Rheumatoid arthritis);
* Known or suspected history of immunosuppression, immune disorders, or immune disorders, including but not limited to invasive opportunistic infections (histoplasmosis, listeriosis, coccidioides, pulmonary cysticercosis disease, aspergillosis), even if the infection has been resolved;
* Any intranasal and/or sinus surgery (including polypectomy) within 6 months before screening;
* Uncontrolled epistaxis occurred within 2 months before screening;
* A history of active pulmonary tuberculosis in the 12 months before screening;
* Infection requiring treatment with systemic antibacterial, antiviral, antifungal, antiparasitic, or antiparasitic agents occurred within 14 days before screening;
* Helminth parasite infection was diagnosed within 24 weeks prior to screening and had not received or failed to respond to standard treatment;
* Leukotriene antagonists/modulators were used while screening (using a stable dose of leukotriene modulator for ≥30 days before screening was acceptable);
* Regular use of decongestants (topical or systemic) before screening, except for short-term use for endoscopy;
* Patients who received any of the following treatments before screening:

  1. Received immunosuppressive therapy within the previous 8 weeks or five half-lives (whichever was longer), (including but not limited to cyclophosphamide, cyclosporine, interferon-γ, azathioprine, methotrexate, mycophenolate mofetil and tacrolimus, etc.);
  2. Received monoclonal antibody therapy within the previous 8 weeks or five half-lives (whichever was longer), (Including but not limited to: benralizumab, mepolizumab, omalizumab, resveratrol, dupilumab, etc.);
  3. Received systemic glucocorticoids within 28 days before the study;
  4. Glucocorticoid-eluting nasal stents were used within 6 months before the study;
  5. Immune globulin or blood products therapy were used within 28 days before the study;
  6. Received or planned to receive live attenuated vaccine within 28 days before or during the study period;
  7. Received allergen specific immunotherapy 6 mouth before screening (if started at 3 mouth before screening, being treated at a stable dose in 1 mouth before visit 1 and not expected to change during study, it would be acceptable);
  8. Join any other clinical trials within 3 months;
* Patients with concurrent asthma had any of the following conditions: forced expiratory volume in the first second (FEV1) ≤ 50% of the expected normal value, or acute exacerbation of asthma within 90 days prior to screening, requiring hospitalization (>24 hours), or taking a daily dose greater than 1000 μg of fluticasone or equivalent inhaled glucocorticoids (ICS);
* Hepatitis B surface Antigen (HBsAg) positive, or Hepatitis B core antibody (HBcAb) positive and Hepatitis B virus deoxyribonucleic acid (HBV-DNA) positive, or anti-hepatitis C virus (Anti-HCV) positive and Hepatitis C virus ribonucleic acid (HCV-RNA) positive, or anti-human Immunodeficiency Virus (Anti-HIV) positive, or anti-treponema pallidum (Anti-TP) positive;
* Any clinically significant abnormal findings, include physical examination, vital signs, 12-lead electrocardiogram, blood biochemistry, blood routine or urine routine, and investigator judged that participating in the trial may put the patient at risk, or may affect the study outcome or hinder the patient's ability to complete the entire study process;
* Lab tests results were abnormal:

  1. White cell count<3.5 x 10^9/L;
  2. Aspartate aminotransferase (AST) > 2.5 x upper limits of normal (ULN);
  3. Alanine aminotransferase (ALT) > 2.5 x ULN;
  4. Total bilirubin > 2 x ULN;
  5. Creatine phosphokinase (CPK)> 2 x ULN;
  6. Creatinine >1.5 x ULN
* Pregnant or lactating women;
* A allergic history or allergic reaction to Mometasone furoate nasal spray (Nasonex®) or any component of TQC2731 injection;
* A history of systemic allergy to any biologic drug (except local injection site reactions);
* The subjects had poor compliance and were judged unable to complete the study;
* Any medical or psychiatric disorder that was considered by the investigator or the sponsor medical reviewer to be likely to affect the safety of the subjects throughout the study or to prevent the subjects from completing the study or interfere with the interpretation of the results; including but not limited to cardiovascular, gastrointestinal, liver, kidney, neurological, musculoskeletal, infectious, endocrine, metabolic, hematological diseases, psychiatric or major limb disorders etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-12-08 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
Nasal Polyp Score (NPS) | Baseline up to 24 weeks
  NPS is the sum of the left and right nostril scores evaluated through nasal endoscopy, with a total score range of 0 to 8. NPS is based on polyp grading, with a score of 0-4 based on polyp grading.

SECONDARY OUTCOMES:
Nasal congestion score (NCS) | Baseline up to 24 weeks
  NCS is determined by the subjects based on the severity of the nasal congestion in the past 24 hours. This score uses a 0-3 classification scale, where 0=no symptoms, 1=mild symptoms, 2=moderate symptoms, and 3=severe symptoms.
Anosmia Score | Baseline up to 24 weeks
  Anosmia Score is evaluated by subjects based on their severity of Anosmia on the day. This score uses a 0-3 classification scale, where 0=no symptoms, 1=mild symptoms, 2=moderate symptoms, and 3=severe symptoms.
Total symptom score (TSS) | Baseline up to 24 weeks
  TSS is the sum of nasal congestion, anosmia, and rhinorrhea (the average of anterior and posterior rhinorrhea), with a score range of 0-9 points. The severity is evaluated by the subject and recorded on the subject diary record card.
Visual analogue scale (VAS) for sinusitis | Baseline up to 24 weeks
  VAS for sinusitis is a questionnaire that subjective evaluation of the overall severity of sinusitis by subjects, with a score range of 0-10 points. The higher the score, the greater the impact of sinusitis on the quality of life of the subjects.
Nasal polyp (NP) surgery time | Baseline up to 32 weeks
  Time to the first nasal polyp (NP) surgery of subjects
Nasal polyp (NP) surgery ratio | Baseline up to 32 weeks
  Ratio of subjects who undergo nasal polyp surgery.
Time of Systemic glucocorticoids (SCS) remedial treatment | Baseline up to 32 weeks
  Time to first use of systemic glucocorticoids (SCS) as remedial treatment of subjects.
Ratio of Systemic glucocorticoids (SCS) treatment | Baseline up to 32 weeks
  Ratio of subjects who using SCS as remedial treatment.
Lund Mackay (LMK) score | Baseline up to 24 weeks
  The LMK score is based on the results of sinus Computed Tomography (CT) scans. Evaluated by researchers, divided into left and right sinus systems, with 0-12 points per side and a total score of 0-24 points.
Incidence of Adverse event (AE) | Baseline up to 32 weeks
  Incidence of AE, serious adverse event (SAE) and abnormal laboratory tests
Severity of AE | Baseline up to 32 weeks
  Severity of AE, serious adverse event (SAE) and abnormal laboratory tests
Peak concentration (Cmax) | Before first administration, 1, 4, 8, 12, 24, 72, 120, 144, 168, 336 hours after first administration; before second, third, fourth and last administration; 1, 4, 8, 12, 24, 72, 168, 336, 672, 1008, 1344, 1992 hours after last administration.
  Maximum plasma drug concentration
Trough concentration (Cmin) | Before first administration, 1, 4, 8, 12, 24, 72, 120, 144, 168, 336 hours after first administration; before second, third, fourth and last administration; 1, 4, 8, 12, 24, 72, 168, 336, 672, 1008, 1344, 1992 hours after last administration.
  Minimum plasma drug concentration
Time to Peak concentration (Tmax) | Before first administration, 1, 4, 8, 12, 24, 72, 120, 144, 168, 336 hours after first administration; before second, third, fourth and last administration; 1, 4, 8, 12, 24, 72, 168, 336, 672, 1008, 1344, 1992 hours after last administration.
  The time when reach maximum plasma drug concentration
Area under the concentration time curve (AUC0-t) | Before first administration, 1, 4, 8, 12, 24, 72, 120, 144, 168, 336 hours after first administration; before second, third, fourth and last administration; 1, 4, 8, 12, 24, 72, 168, 336, 672, 1008, 1344, 1992 hours after last administration.
  The area enclosed by the plasma concentration curve to the timeline
Maximum plasma concentration at steady state (Css-max) | Before first administration, 1, 4, 8, 12, 24, 72, 120, 144, 168, 336 hours after first administration; before second, third, fourth and last administration; 1, 4, 8, 12, 24, 72, 168, 336, 672, 1008, 1344, 1992 hours after last administration.
  The maximum plasma concentration after stabilization
Minimum plasma concentration at steady state (Css-min) | Before first administration, 1, 4, 8, 12, 24, 72, 120, 144, 168, 336 hours after first administration; before second, third, fourth and last administration; 1, 4, 8, 12, 24, 72, 168, 336, 672, 1008, 1344, 1992 hours after last administration.
  The minimum plasma concentration after stabilization
Plasma concentration at steady state (Css-av) | Before first administration, 1, 4, 8, 12, 24, 72, 120, 144, 168, 336 hours after first administration; before second, third, fourth and last administration; 1, 4, 8, 12, 24, 72, 168, 336, 672, 1008, 1344, 1992 hours after last administration.
  The plasma concentration at which the rate of administration and rate of elimination are in equilibrium.
Time to Peak concentration at steady state (Tss-max) | Before first administration, 1, 4, 8, 12, 24, 72, 120, 144, 168, 336 hours after first administration; before second, third, fourth and last administration; 1, 4, 8, 12, 24, 72, 168, 336, 672, 1008, 1344, 1992 hours after last administration.
  The time when maximum plasma drug concentration at steady state.
Area under the concentration time curve (AUC0-t) at steady state | Before first administration, 1, 4, 8, 12, 24, 72, 120, 144, 168, 336 hours after first administration; before second, third, fourth and last administration; 1, 4, 8, 12, 24, 72, 168, 336, 672, 1008, 1344, 1992 hours after last administration.
  The area enclosed by the plasma concentration curve to the timeline at steady state.
Half life (t1/2) | Before first administration, 1, 4, 8, 12, 24, 72, 120, 144, 168, 336 hours after first administration; before second, third, fourth and last administration; 1, 4, 8, 12, 24, 72, 168, 336, 672, 1008, 1344, 1992 hours after last administration.
  The time taken for the plasma concentration to be reduced by half.
Apparent volume distribution (Vd/F) | Before first administration, 1, 4, 8, 12, 24, 72, 120, 144, 168, 336 hours after first administration; before second, third, fourth and last administration; 1, 4, 8, 12, 24, 72, 168, 336, 672, 1008, 1344, 1992 hours after last administration.
  It refers to the ratio between the body drug amount and the blood drug concentration after the drug has reached dynamic equilibrium in the body.
Plasma clearance (CL/F) | Before first administration, 1, 4, 8, 12, 24, 72, 120, 144, 168, 336 hours after first administration; before second, third, fourth and last administration; 1, 4, 8, 12, 24, 72, 168, 336, 672, 1008, 1344, 1992 hours after last administration.
  The volume of plasma cleared of drug per unit time.
Anti-drug antibody (ADA) | Within 1 hour before administration on Day 1, Day 169, Day 224, during withdrawal
  Incidence and their titers of Anti-drug antibody (ADA)
Neutralizing antibody (Nab) | Within 1 hour before administration on Day 1, Day 169, Day 224, during withdrawal
  Incidence and their titers of Neutralizing antibody (Nab)

CONTACTS AND LOCATIONS:
Locations (16):
- China (16):
  - The First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - ZhuJiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Jieyang People's Hospital, Jieyang, Guangdong
  - The Fifth Affiliated Hospital Sun Yat-sen University, Zhuhai, Guangdong
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Affiliated Zhongshan Hospital Of Dalian University, Dalian, Liaoning
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Weifang Second People's Hospital, Weifang, Shandong
  - Eye & ENT Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Chengdu Second People's Hospital, Chengdu, Sichuan
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang Uygur Autonomous Region